CLINICAL TRIAL: NCT04095416
Title: Compression Wraps as Adjuvant Therapy in the Management of Acute Systolic Heart Failure (CATAS-HF)
Brief Title: Compression Wraps as Adjuvant Therapy in Management of Acute Systolic Heart Failure
Acronym: CATAS-HF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: challenges in recruitment due to covid-19
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Joseph Miller, MD, Emergency Medicine, Internal Medicine Physician, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CATASHFtrial2019
Record Dates: First submitted 2019-08-13; First posted 2019-09-19 (Actual); Results first posted 2022-02-24 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Heart Failure; With Decompensation
Keywords: Compression wraps; heart failure; systolic; edema; wrap
MeSH Terms: conditions — Heart Failure; Systolic Murmurs; Edema

STUDY DESIGN:
Intervention Model Description: Two arms, one interventional group and one control. Interventional group receives compression wraps and standard medical care, control group only receives standard medical care
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Intervention (Experimental): Bilateral lower extremity ACE compression wraps in addition to standard medical care
  Interventions: Device: ACE compression wrap
- Control (No Intervention): Standard medical care

INTERVENTIONS:
Device: ACE compression wrap — Bilateral lower extremity ACE compression wraps
  Arms: Intervention

SUMMARY:
There will be two populations in this study: control group, and intervention group. These groups will undergo propensity matching to account for confounders and minimize selection bias. 120 patients will be enrolled, 60 to each population. The objective of this study is: assess the utility of lower extremity compression wraps as adjuvant therapy in inpatient management of acute systolic heart failure

The control group will consist of patients admitted to I5 Cardiology for management of acute systolic heart failure with intravenous diuresis and standard medical therapy, meeting inclusion criteria. Information will be gathered through observational prospective data analysis from Epic EMR, and will include daily diuretic type and dose required, daily urine output, daily creatinine, total days of admission, daily and pre-discharge weight, admission BNP, and pre-discharge BNP.

The intervention group will consist of patients admitted to I5 Cardiology meeting inclusion criteria and being managed with standard medical therapy. This group will receive additional therapy using bilateral lower extremity compression wraps applied by nursing staff per pre-set protocol, and will receive education on the use of compression wraps. Patients will be instructed to wear the compression wraps for the entirety of the time they are undergoing intravenous diuresis, with pauses in care as needed for hygiene and symptom relief purposes. During the time of compression wrap application, the following data will be collected: urine output, daily weights, daily creatinine, daily and total dose and type of intravenous diuretic used. Prior to discharge, a BNP will be obtained.

Endpoints (including percentage of weight reduction, total urine output achieved with diuresis, total dose requirement and type of intravenous diuresis, total days of intravenous diuresis, days to discharge, discharge BNP, and percent reduction from admission BNP) will then be compared to assess the utility of adding lower extremity compression wraps to inpatient management of acute systolic heart failure.

DETAILED DESCRIPTION:
There will be two populations in this study: control group, and intervention group. 120 patients will be enrolled, 60 to group, randomized in 1:1 fashion. The control group will consist of patients admitted to I5 Cardiology for management of acute systolic heart failure with intravenous diuresis and standard medical therapy, meeting inclusion criteria. Information will be gathered through observational prospective data analysis from Epic EMR, and will include daily diuretic type and dose required, daily urine output, daily creatinine, total days of admission, daily and pre-discharge weight, admission BNP, and pre-discharge BNP. The intervention group will consist of patients admitted to I5 Cardiology meeting inclusion criteria and being managed with standard medical therapy. This group will receive additional therapy using bilateral lower extremity compression wraps applied by nursing staff per pre-set protocol, and will receive education on the use of compression wraps. Patients will be instructed to wear the compression wraps for the entirety of the time they are undergoing intravenous diuresis, with pauses in care as needed for hygiene and symptom relief purposes. During the time of compression wrap application, the following data will be collected: urine output, daily weights, daily creatinine, daily and total dose and type of intravenous diuretic used. Prior to discharge, a BNP will be obtained. Endpoints (including percentage of weight reduction, total urine output achieved with diuresis, total dose requirement and type of intravenous diuresis, total days of intravenous diuresis, days to discharge, discharge BNP, and percent reduction from admission BNP) will then be compared to assess the utility of adding lower extremity compression wraps to inpatient management of acute systolic heart failure.

ELIGIBILITY:
Inclusion Criteria:

* age greater than 18 and less than 85 years of age
* admitted to I5 with Acute Systolic Heart Failure with an ejection fraction of less than 50% as determined by echocardiogram within 6 months
* requiring inpatient management with intravenous diuresis.
* diagnosis of acute systolic heart failure, of any underlying etiology
* at least 2+ pitting edema (or documented lower extremity pitting edema of at least moderate or significant severity) on primary assessment.

Exclusion Criteria:

* cannot tolerate IV diuresis
* who cannot wear or tolerate lower extremity compression stockings or wraps
* ESRD
* peripheral neuropathy
* ejection fraction greater than 50% as evaluated by echocardiogram within 6 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2021-01-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment terminated early due to COVID-19 pandemic
Groups:
- Intervention: Bilateral lower extremity compression wraps in addition to standard medical care
  Compression wrap: Bilateral lower extremity compression wraps applied by trained research team
Period: Overall Study
Arm/Group | Intervention | Control
Started | 13 | 19
Completed | 10 | 19
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention: Adult patients age 18 years or older with a history of chronic heart failure (functional class II, III, or IV) with a left ventricular ejection fraction of 40% or less as determined by echocardiography within 6 months of evaluation, were eligible for enrollment in the trial. Final inclusion criteria required admission to the telemetry unit for intravenous (IV) diuretic therapy in the management of acute decompensated heart failure, and presence of lower extremity pitting edema on physical examination.
  Bilateral lower extremity compression wraps in addition to standard medical care
  Compression wrap: Bilateral lower extremity compression wraps applied by trained research team
- Control: Adult patients age 18 years or older with a history of chronic heart failure (functional class II, III, or IV) with a left ventricular ejection fraction of 40% or less as determined by echocardiography within 6 months of evaluation, were eligible for enrollment in the trial. Final inclusion criteria required admission to the telemetry unit for intravenous (IV) diuretic therapy in the management of acute decompensated heart failure, and presence of lower extremity pitting edema on physical examination.
  Standard medical care
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 10 | 19 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 8 | 12
  >=65 years | 6 | 11 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (16) | 64 (12) | 64 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 7 | 15 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 12 | 18
  White | 4 | 7 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Admission weight [Mean (Standard Deviation); unit: kg] | 98.3 (30.9) | 91.2 (21.3) | 93.7 (24.7)
Admission BNP [Mean (Standard Deviation); unit: pg/mL] | 2279 (1613) | 1997 (1296) | 2095 (1391)
Ejection fraction, baseline [Mean (Standard Deviation); unit: %] | 32 (10) | 26 (9) | 28 (10)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Readmission Within 30-days
Description: Assess rate of 30-day readmission of patients enrolled in study
Time Frame: 30 days from hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 10 | 19
Participants | 2 | 5

2. Primary Outcome: Total Length of Hospital Stay
Description: Assess the length of hospitalization, controlling for variables
Time Frame: From admission to hospital discharge, up to 30 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention | Control
Number analyzed (Participants) | 10 | 19
days | 4.6 (2.6) | 7.4 (3.9)

3. Primary Outcome: Days on IV Diuretic Therapy
Description: Assess the number of days from start of IV diuresis to transition to PO diuresis
Time Frame: From admission to hospital discharge, up to 30 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention | Control
Number analyzed (Participants) | 10 | 19
days | 4.2 (3.1) | 5.0 (1.8)

4. Secondary Outcome: Average Percentage of BNP Change
Description: Assess the average percent of BNP reduction of intervention vs control groups
Time Frame: From admission to hospital discharge, up to 30 days
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Intervention | Control
Number analyzed (Participants) | 10 | 19
% change | -38.5 (22.8) | -38.2 (57.6)

5. Secondary Outcome: Average Pre-discharge BNP
Description: Assess the average pre-discharge BNP of intervention vs control groups
Time Frame: From admission to hospital discharge, up to 30 days
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Intervention | Control
Number analyzed (Participants) | 10 | 19
pg/mL | 1404 (1441) | 1238 (896)

6. Secondary Outcome: Net Intake/Output of Fluids During Hospitalization
Description: Assess the net intake/output across the hospitalization of intervention vs control groups, obtained through nursing documentation of fluid intake and output recorded daily during the hospitalization
Time Frame: From admission to hospital discharge, up to 30 days
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Intervention | Control
Number analyzed (Participants) | 10 | 19
L | -8.13 (8.05) | -7.08 (6.21)

7. Secondary Outcome: IV Diuretic Infusion Used
Description: Assess the use of IV diuretic in intervention vs control groups
Time Frame: From admission to hospital discharge, up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 10 | 19
Participants | 0 | 7

8. Secondary Outcome: Average Percentage of Weight Change During Hospitalization
Description: Assess the average percent of weight reduction of intervention vs control groups
Time Frame: From admission to hospital discharge, up to 30 days
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Intervention | Control
Number analyzed (Participants) | 10 | 19
% change | -7.2 (6.1) | -5.7 (5.2)

9. Secondary Outcome: AKI During Hospitalization
Description: Development of acute kidney injury during hospitalization
Time Frame: From admission to hospital discharge, up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 10 | 19
Participants | 1 | 13

ADVERSE EVENTS:
Time Frame: Up to 30 days after discharge
Description: Does not differ from clinicaltrials.gov definition
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/19
Other Adverse Events (participants affected / at risk) | 0/10 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-01): https://cdn.clinicaltrials.gov/large-docs/16/NCT04095416/Prot_SAP_002.pdf
  • Informed Consent Form (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/16/NCT04095416/ICF_003.pdf